CLINICAL TRIAL: NCT05052242
Title: Evaluation of Ocular Biometry in Primary Angle-closure Disease With Two Swept Source Optical Coherence Tomography Devices
Brief Title: Evaluation of Ocular Biometry in PACD With Two Swept Source Optical Coherence Tomography Devices
Status: Completed | Type: Observational
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Other Study IDs: Rajavithi hospital
Record Dates: First submitted 2021-09-03; First posted 2021-09-22 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Primary Angle Closure Glaucoma
Keywords: Ocular biometry; swept source OCT; agreement
MeSH Terms: conditions — Glaucoma, Angle-Closure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- one group compared two measurement methods: one group compared two measurement methods
  Interventions: Diagnostic Test: primary angle closure disease

INTERVENTIONS:
Diagnostic Test: primary angle closure disease — 2 swept source OCT biometers, IOL Master700 and Anterion

SUMMARY:
Purpose: To investigate agreement between 2 swept source OCT biometers, IOL M.aster700 and Anterion, in various ocular biometry and intraocular lens (IOL) calculations of primary angle-closure disease (PACD).

Methods: This was a prospective study conducted in a tertiary eye care centre involving biometric measurements obtained with 2 devices in phakic eye with diagnosis of PACD. Mean difference and intraclass correlation coefficient (ICC) with confidence limits were assessed, and calculations of estimated residual refraction of the IOL were analysed using Barrett's formula.

DETAILED DESCRIPTION:
Primary angle-closure disease (PACD) is the leading cause of blindness worldwide. PACD is an anatomic disorder, typically of relatively small eye with shallow anterior chamber depth (ACD), thick lens, shorter axial length (AL), small corneal curvature, and relatively anterior lens position. Pupillary block, plateau iris and phacomorphic mechanisms play major roles in the pathophysiology of the disease, and pupillary block is thought to be the most common causal mechanism.

For decades, phacoemulsification and intraocular lens implantation (PEI) has been proposed for initial management of PACD.4 PEI relieves pupillary block, deepening ACD and widening irido-corneal angle.

Biometry is essential in evaluating ocular dimensions and calculating IOL power in PACD, and ocular biometers have been evolving in recent years. Optical coherence tomography (OCT) includes partial coherence interferometry (PCI), and swept source OCT (SS-OCT) is in general use in clinical practice. The agreement of the calculations of these devices has been studied by many investigators; however, research into their agreement in PACD patients has been sparse so far. A newer SS-OCT, Anterion, is now available and its performance needs to be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were age > 40 years old
* phakic eye
* diagnosis of PACD, including primary angle-closure suspect (PACS), primary angle-closure (PAC) and primary angle-closure glaucoma (PACG) as classified by Foster et al

Exclusion Criteria:

* patients who had opaque optical media
* dense cataract
* anterior and/or posterior segment diseases such as advanced pterygium, diabetic retinopathy, or maculopathy
* Participants who had previous history of ocular trauma, ocular surgery

Ages: 40 Years to 77 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: participants from the glaucoma clinic at Rajavithi Hospital, Bangkok, Thailand. between May and December 2020
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-09-03 (Actual)

PRIMARY OUTCOMES:
Intraclass correlation coefficient of IOL power calculation | 30 minutes per person
  agreement between 2 swept source OCT biometers, IOL Master700 and Anterion, in intraocular lens (IOL) calculations
Intraclass correlation coefficient of various ocular biometry | 30 minutes per person
  agreement between 2 swept source OCT biometers, IOL Master700 and Anterion, in various ocular biometry( ACD, AL, LT, K1, K2, WTW)

CONTACTS AND LOCATIONS:
Overall Officials: Somporn Chantra, MD, Principal Investigator — Department of Medical Services Ministry of Public Health of Thailand
Locations (1):
- Somporn Chantra, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No